CLINICAL TRIAL: NCT05116852
Title: Community and Familial Impacts of the Opioid Crisis
Status: Completed | Type: Observational
Sponsor: Cambridge Health Alliance (Other)
Collaborators: The Sandra and Arnold Gold Humanism Research Fund (Unknown)
Responsible Party: Principal Investigator, Zev Schuman Olivier, Assistant Professor, Psychiatry, Cambridge Health Alliance
Other Study IDs: CHA-IRB-20-21-7
Record Dates: First submitted 2021-10-13; First posted 2021-11-11 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Bereavement; Overdose of Opiate
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Both grieving a loved one to opioid-related death and have an actively using loved one: These individuals will complete the study survey for their designated experience both supporting a loved one in treatment for Opioid Use Disorder, and having lost a loved one to opioid-related death.
  Interventions: Other: Survey
- Individuals supporting a loved one in treatment for Opioid Use Disorder: These individuals will complete the study survey for their designated experience supporting a loved one in treatment for Opioid Use Disorder.
  Interventions: Other: Survey
- Individuals grieving a loved one to opioid-related death: These individuals will complete the study survey for their designated experience losing a loved one to opioid-related death.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — All study participants will be asked to complete two surveys relevant to their personal experience either losing a loved one to opioid-related death, supporting a loved on in recovery for Opioid Use Disorder, or both.

SUMMARY:
This study aims to analyze the needs of those who have lost a loved one to opioid-related death and/or those currently supporting a loved one in treatment for Opioid Use Disorder. Mental health status related to the death or support of a loved one will be assessed through a survey and through the use of several modules of the CAT-MH (computerized adaptive testing-mental health suite) questionnaire.

DETAILED DESCRIPTION:
This study aims to establish the level of needs in the community among those who have lost loved ones to opioid overdose and/or currently support those in opioid addiction recovery. This study aims to analyze the needs of those who have lost a loved one to opioid-related death and/or those currently supporting a loved one in treatment for Opioid Use Disorder. The study will evaluate the mental health status for each study participant through a primary survey as well as current participant mental health status through the use of several modules of the CAT-MH adaptive testing questionnaire. CAT-MH will be used to rapidly measure severity levels of depression, anxiety, and substance use risk after participants complete the primary survey. The primary survey assesses the immediate impact of overdose death by a loved one and recognition of the onset of opioid addiction in the years after the event on family and community members. The primary survey will compare the impact of loss and/or recovery support on mental health and substance use at specified time points before and after the loss and/or an individual finding out about a loved one's opioid addiction. The primary survey will also evaluate attitudes in this population about mindfulness and self-compassion skills training, openness to technology and various treatment options, current and past levels of depression, anxiety and grief, as well as thematic areas of need specific to those who have lost a loved one to opioid overdose and/or currently support a loved one in opioid addiction recovery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+, inclusive, who are competent, wish to participate and willing to provide informed consent
* Willing and able to participate in completing the surveys using the internet on via smartphone as requested
* Identify in one of the 3 groups: (a) Adults who have lost a direct relative or friend to opioid overdose or opioid-related death prior to taking the survey; (2) Adults who are currently supporting a loved one with active opioid addiction; (3) Adults who have lost a direct relative or friend to opioid overdose or opioid related death at least six months prior to survey participation and also currently support a loved one in active addiction recovery.

Exclusion Criteria:

* Inability to complete the survey
* Inability to speak, read, and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected by an email send both to collaborating organizations that provide peer support for those with addiction-related overdose and to healthcare systems that provide care for people with OUD to share with people in their communities who may have lost a loved one to opioid-related death.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Establish the percentage of adults who have lost a loved one to opioid overdose who had increased substance use in the year after their loss. | Day 1
  This self-report aim will be assessed via participant survey response asking for recollection of substance use before and after the loss.

SECONDARY OUTCOMES:
Establish the percentage of adults who have lost a loved one to opioid overdose who received mental health treatment in the year after their loss. | Day 1
  This self-report aim will be assessed via participant survey response asking for recollection of mental health treatment before and after the loss.
Compare the level of negative impact on substance use and mental health status in the year after loss due to overdose with the impact on substance use and mental health in the year after becoming aware of a child's opioid addiction. | Day 1
  This aim will be assessed via participant survey response between cohorts
Prolonged Grief | Day 1
  Aa version of the prolonged grief (PG-13) scale will be used to assess presence of prolonged grief after date of loss event.

OTHER OUTCOMES:
Depression | Day 1
  This aim will be assessed via CAT-MH's CAT-DI adaptive test (computerized adaptive testing-mental health suite for depression).
Establish the percentage of adults who have lost a loved one to opioid overdose who had worsening eating disorders, OCD (Obsessive-compulsive disorder), or problematic sexual behaviors in the year after their loss. | Day 1
  This aim will be assessed via participant survey self-report responses.
Anxiety | Day 1
  This aim will be assessed via CAT-MH's CAT-Anxiety adaptive test
PTSD symptoms | Day 1
  This aim will be assessed via CAT-MH's CAT-PTSD adaptive test
Establish the percentage of adults who have lost a loved one to opioid overdose who had worsening depression in the year after their loss. | Day 1
  This self-report aim will be assessed via participant survey response asking for recollection of depression symptoms before and after the loss.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided